CLINICAL TRIAL: NCT07134686
Title: Implementation of a Joint Pulmonologist and ENT Consultation in the Care Pathway of Patients Suffering From Asthma and Chronic Rhinosinusitis With Nasal Polyposis: Effectiveness Compared With Consultations by Specialty (CON-PO Study).
Acronym: CON-PO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-A02003-44
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Asthma; Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Keywords: Asthma; Care pathway; Chronic Rhinosinusitis with Nasal Polyps (CRSwNP)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint consultation (Experimental): Multi-disciplinary consultation with a pulmonologist and ENT specialist at the baseline visit
  Interventions: Other: Joint consultation; Procedure: Mucus sampling; Procedure: Nasal brushing
- Separate consultations (Active Comparator): Separate consultations with a pulmonologist and ENT specialist at the baseline visit as standard care
  Interventions: Procedure: Mucus sampling; Procedure: Nasal brushing

INTERVENTIONS:
Other: Joint consultation — Joint consultation with pneumologist and ENT at baseline.
  Arms: Joint consultation
Procedure: Mucus sampling — Mucus sampling at baseline and one year follow-up
Procedure: Nasal brushing — Nasal brushing at baseline and one year follow-up

SUMMARY:
Asthma affects the lower respiratory tract (bronchi), whereas chronic rhinosinusitis with nasal polyposis (CRSwNP) involves the upper airways. Despite this anatomical distinction, the upper and lower airways form a continuous respiratory tract and share common pathophysiological mechanisms. Consequently, asthma and CRSwNP frequently coexist, and several therapeutic strategies are effective for both conditions.

Given these overlaps, we hypothesize that a multidisciplinary consultation involving both a pulmonologist and an ENT specialist could be more effective than separate consultations for patient care. We also believe that this innovative organization that would benefit the healthcare system.

To test this hypothesis, we are conducting a study whose primary objective is to assess whether joint consultations lead to a reduction in oral corticosteroid need over the year following the initial consultation, by enabling more personalized treatment strategies.

Secondary outcomes will include the frequency of asthma exacerbations, frequency of ENT-related events, respiratory symptoms, quality of life, and healthcare ressources utilization.

We will compare outcomes between two patient groups: one receiving joint consultation from both specialists, and the other managed through standard, separate consultations as per current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older;
* With a diagnosis of asthma;
* With a diagnosis of chronic rhinosinusitis with nasal polyposis;
* Whose asthma and/or chronic rhinosinusitis is/are not controlled according to SNOT-22 and ACQ-6 scores;
* Having used systemic corticosteroids in the previous year to treat symptoms related to one of these conditions at least;

Exclusion Criteria:

* Patient in a period of exclusion from another research protocol at the time of consent signature;
* Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code (adult patients under guardianship or curatorship, patients deprived of their liberty, pregnant or breast-feeding women);
* Patients who do not read and/or understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of joint ENT and pulmonologist consultation on relative change in cumulative annual dose of oral corticosteroids from the year before Baseline to the year between Baseline and 12 months visit. | From the year before Baseline to the 12 months visit.
  Self reported cumulative annual dose of oral corticosteroids.

SECONDARY OUTCOMES:
Reduction of asthma exacerbations frequency. Relative change from the year before Baseline to the year between baseline and 12 months visit in number of asthma exacerbations. | From the year before Baseline to the 12 months visit.
  self-reported number of asthma exacerbations
Reduction of ENT events frequency. Relative change from the year before baseline to the year between baseline and 12 month visit in number of ENT events. | From the year before Baseline to the 12 months visit.
  Self reported number of ENT events
Improvement of asthma control. Relative change from baseline to 12 months visit in ACQ-6 score | Baseline and 12 months visit.
  Self-administered questionnaire
Improvement of chronic rhinosinusitis with nasal polyposis control . Relative change from baseline to 12 months visit in SNOT-22 score | Baseline and 12 months visit.
  Self-administered questionnaire
Reduction in endoscopic polyp score. Relative change from baseline to 12 months visit in the polyp endoscopic score (mean of measures of both nostrils) | Baseline and 12 months visit.
  Evaluated with nasal endoscopy
Improvement of patient's quality of life. Relative change from baseline to 12 months visit in EQ-5D-5L score | Baseline and 12 months visit.
  Self-administered questionnaire
Reduction of healthcare ressource use . Relative change from baseline to 12 months visit in number of consultations with a specialist, general practitionner, emergency visits and hospitalizations | From Baseline to the 12 months visit
  Self-reported number of consultations with a specialist, general practicionner, emergency visits and hospitalizations